CLINICAL TRIAL: NCT01216215
Title: Novel Gentic Variations Contributing to Asthma Susceptability in Saudi Arabia
Status: Completed | Type: Observational
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Saleh Zaid Al-Muhsen, Associate Professor, King Saud University
Other Study IDs: SaudiGenAsthma; King saud University (Other: King saud University)
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Collection of Clinical Data That Will be Used in This Study and Will Form a Data Bank for Asthma in Saudi Arabia; Identify Known and NOVEL Genetic Risk Factors Contributing to Asthma Susceptibility; Study the Mechanistic Roles of the Genetic Variants Within Major Asthma Susceptibility Genes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Asthmatic sporadic and familial
- Control subjects spradic and familial

SUMMARY:
Research Problem Asthma is one of the most common chronic diseases in the world that affects approximately 300 million individuals worldwide. It is characterized by airway inflammation and bronchoconstriction leading to airflow obstruction, however, the triggering factors behind asthma development remains to be elucidated. Genetic risk factors have been suggested to play a central role in asthma development. Twin studies supported a strong genetic component to asthma, especially childhood asthma, with heritability estimates suggesting that 48-70% of asthma risk is attributed to genetic risk factors. Suggestive susceptibility genes have been identified in European and American populations but not yet in the Middle East including Saudi Arabia. Identified genes whether they are polymorphic variants of genes encoding known pathophysiological molecules or novel genes identified by linkage or genome-wide association studies (GWAS) are inconsistent in different populations thereby adding to the need to undertake genetic studies on different ethnic populations and in different countries. Here, the investigators hypothesize that polymorphic variation of novel susceptibility genes form a major risk factor for asthma development, response to treatment and progression in the Saudi population with strong diagnostic, prognostic and therapeutic implications.

Research Significance Since the manifestation of complex inflammatory disorders with strong heritability is complex involving genetic and environmental interaction, each ethnically distinct population must be examined to know whether gene-disease association exists in that population. The objectives of this proposal are to discover novel asthma susceptibility genes in the Saudi population. A better understanding of the genetic mechanisms of asthma will enhance our knowledge of its pathophysiology. Asthmatic patients with distinct genotypes respond differently to asthma medications. Therefore, improvements in diagnostics and pharmacogenetics may be the first clinical developments of these extensive studies. This embraces the concept of asthma subphenotypes and stratified medicine where interventions are targeted at those individuals who will best benefit from them with minimal side effects. Physicians looking after asthmatic patients will be able to provide better medical service tailored to those patients, as well as to identify Saudi people at high risk for the development of asthma, especially the more severe forms of the disease.

Research Objectives The main objective of our proposal is to identify known and novel asthma susceptibility genes in the Saudi population and to investigate their interaction with clinical, environmental, and inflammatory factors contributing to asthma pathophysiology.

Research Methodology In this proposal, the investigators will investigate the genetic factors contributing to asthma susceptibility by determining in Saudi population, the presence of single nucleotide polymorphisms (SNPs) that have been previously reported from linkage and GWAS in other populations. Whole genome DNA will also be scanned for novel SNPs of selected "asthma genes" using microarrays. This will enable us to identify new SNPs that contribute to the risk of asthma specifically in the Saudi population. In addition, the investigators will cross-reference all genetic and immunological parameters with the corresponding clinical data in order to elucidate the impact of certain genes, or their products (e.g. cytokines), on the clinical manifestation of asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with documented clinical history of asthma for a period of at least 6 months prior to study entry (and a minimum of one clinic follow-up visit since initial diagnosis)
2. Willing to provide written informed consent and in the judgment of the investigator, individuals who are able to understand the informed consent process.
3. Subjects with documented clinical history (in preceding 12 months) of airway reversibility of at least 12% based on Forced Expiratory Volume (FEV1), measured pre and post inhalation of a β-2 agonist (2 puffs of albuterol using a measured dose inhaler with spacer) OR
4. Individuals demonstrating airway 12% reversibility during recruitment testing and asthmatic symptoms, but with no prior history of asthma and not on an asthma treatment plan, can be recruited as affected individuals if in the opinion of the investigator the individuals are truly asthmatic and have no confounding factors that could explain the reversibility and symptoms.

7. Individuals with strong history of asthma but with waning, or no current symptoms may be included in the study if their asthma was well controlled using an asthma medication. Principal investigator must verify or know the clinical history of an individual before accepting him as an asthmatic individual.

8. Individuals with positive history of asthma but no asthma medication usage and with family history of asthma should be considered for inclusion as cases in the study only if other family members are being recruited.

9. Able to perform Spirometry/FEV1 correctly (only for those above 7years).

Exclusion Criteria:

1. Age < 3 years
2. Smoking for 20 years, 1 pack/day or more.
3. Congestive heart failure.
4. COPD.
5. Chronic lung disease other than asthma and COPD.
6. Bronchiectasis.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is a multi-center observational study. Asthmatic patients attending major hospitals in Riyadh with clear and well defined inclusion criteria (see below for details, Appendix I) will be recruited. We anticipate recruiting 1000 asthmatic patients and comparable number of control subjects. The controls will be recruited from people attending blood bank for donation or other patients attending different clinics with history excluding atopic diseases and asthma. Ethical approval for this study will be obtained from CMRC ethical committee of the KKUH as well as other involved centers
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2010-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
IL-4 receptor alpha and STAT6 single nucleotide polymorphisms are associated with increased risk of asthma in a Saudi Arabian population. | 2 years
  IL-4Rα rs1805010 and rs1801275 SNPs have been found to be significantly associated with asthma susceptibility in different ethnic groups; some STAT6 SNPs, including rs324011 and rs324015, have also been associated with asthma predisposition and/or IgE levels. Risk evaluations of IL-4Rα and STAT6 SNPs in association with asthma have never been evaluated in Saudi Arabian populations. Methods: Saudi Arabian patients with documented history of severe asthma (n=190) and healthy subjects (n=194) were recruited. Allelic and genotype association to asthma was assessed for IL-4Rα and STAT6 polymorphisms using nucleotide sequencing. Results: The IL4Rα rs1801275 SNP A/G-G/G genotypes, but not the A/A genotype, were significantly associated with asthma predisposition (OR=0.47; 95% CI=0.31-0.72; P<0.001*; dominant model); Similarly, for STAT6 rs324011, odds were significantly higher that homozygous T/T genotype could be associated with asthma.

CONTACTS AND LOCATIONS:
Locations (1):
- King Khalid University Hospital, College of Medicne, King saud University, Riyadh, Central, Saudi Arabia

REFERENCES:
- [Result] Al-Khayyat AI, Al-Anazi M, Warsy A, Vazquez-Tello A, Alamri AM, Halwani R, Alangari A, Al-Frayh A, Hamid Q, Al-Muhsen S. T1 and T2 ADAM33 single nucleotide polymorphisms and the risk of childhood asthma in a Saudi Arabian population: a pilot study. Ann Saudi Med. 2012 Sep-Oct;32(5):479-86. doi: 10.5144/0256-4947.2012.479. PMID 22871616
- See also: Recently published paper. To appear on Pubmed soon. — http://www.thoracicmedicine.org/article.asp?issn=1817-1737;year=2014;volume=9;issue=2;spage=81;epage=86;aulast=Al-Muhsen